CLINICAL TRIAL: NCT06303063
Title: A Prospective, Multicenter, Randomized Controlled Trial to Evaluate the Safety and Effectiveness of the SINOMED IAS for the Treatment of Intracranial Aneurysms
Brief Title: Compare the Safety and Effectiveness of Two Different Kinds of Stent System in Intracranial Aneurysms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinomed Neurovita Technology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNSC-IAS-202301
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Intracranial Aneurysm
Keywords: wide-necked cerebral aneurysms; Brain Aneurysm; Cerebral Aneurysm; Stent
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SINOMED IAS Stent System (Experimental): The SINOMED IAS Stent System is intended for use with occlusive devices in the treatment of intracranial aneurysms.
  Interventions: Device: SINOMED IAS Stent System
- Neuroform Atlas Stent System (Active Comparator): The Neuroform Atlas Stent System is intended for use with occlusive devices in the treatment of intracranial aneurysms.
  Interventions: Device: Neuroform Atlas Stent System

INTERVENTIONS:
Device: SINOMED IAS Stent System — Stent-assisted coiling (SAC) of intracranial aneurysms paved the way for endovascular coiling of wide-neck aneurysms, improving rates of aneurysm obliteration and recurrence.
  Arms: SINOMED IAS Stent System
Device: Neuroform Atlas Stent System — Stent-assisted coiling (SAC) of intracranial aneurysms paved the way for endovascular coiling of wide-neck aneurysms, improving rates of aneurysm obliteration and recurrence.
  Arms: Neuroform Atlas Stent System

SUMMARY:
The primary objective of this trial is to evaluate the safety and efficacy of SINOMED IAS in patients with intracranial aneurysms.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, 1:1 randomized clinical trial to evaluate the safety and efficacy of stent system in the treatment of intracranial aneurysms. A total of 204 patients are planned to be included. The primary endpoint is the incidence of success aneurysm occlusion at 6-month post procedure. All patients will have clinical follow-up during intraoperative, 30 days, 6 months, 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years to 80 years.
2. Wide-necked (Wide-necked is defined as width ≥ 4 mm or a dome-to-neck ratio < 2), saccular, intracranial aneurysms arising from a parent vessel with a diameter of ≥ 2.5 mm and ≤ 5mm.
3. Modified Rankin Scale (mRS) ≤ 2.
4. Subject understands the nature of the procedure, provides voluntary written informed consent prior to the treatment, and is willing to comply with specified follow-up evaluation.
5. The investigators judged the use of stent-assisted coil embolization to be appropriate for the treatment of intracranial aneurysm.

Exclusion Criteria:

1. Target aneurysm is an aneurysm requiring staged procedure.
2. Target aneurysm that has been previously treated with vascular embolization or surgery.
3. Target aneurysms are fusiform aneurysms, dissecting aneurysms, pseudoaneurysms, blood blister-like aneurysms, infected aneurysms, aneurysms associated with arteriovenous malformations.
4. Hospitalized surgical treatment within 30 days before operation, or planned hospitalized surgical treatment within 6 months after surgery.
5. Acutely ruptured aneurysm within 14 days of enrollment.
6. Hunt and Hess (H&H) scale ≥3.
7. Subject who had Moyamoya disease, arteriovenous malformations, arteriovenous fistulae, intracranial tumors, or intracranial mass lated to target aneurysms.
8. Severe stenosis or tortuosity of intracranial arteries or anatomical anomalies that make it difficult to reach the site of the lesion with device.
9. Platelet count <50*103/mm3 (50*109/L) or any known coagulation deficiency, or International normalized ratio (INR)>3.0.
10. Known hypersensitivity/allergies or contraindication to contrast media, stent components, antiplatelets, anticoagulants.
11. Life expectancy < 1 year, and unable to complete the required follow-ups;
12. Female who was pregnant or breastfeeding, women/men planning to havve children in the next year.
13. Currently enrolled in another investigational device or drug study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Success aneurysm occlusion at 6 month post procedure | 6 months post procedure
  The Raymond-Roy occlusion classification (RROC) is an angiographic classification scheme for grading the occlusion of flow diverter treated cerebral aneurysms (class I: complete obliteration, class II: residual neck, class III: residual aneurysm). Higher class represent a worse outcome. The percentage of Success aneurysm occlusion in which class 1 or 2 is achieved on the Raymond Scale at the 6 months follow-up angiographic assessments will be evaluated.

SECONDARY OUTCOMES:
Technical success | Intra-procedure
  Technical success defined as stable stent placement with complete coverage across the aneurysm neck and parent artery patency.
Success aneurysm occlusion immediately after the procedure | Immediately after the procedure
  The percentage of aneurysms in which class 1 or 2 is achieved on the Raymond Scale immediately post-procedure angiographic assessments, will be evaluated.
Complete aneurysm occlusion without significant parent artery stenosis (≤50%) or retreatment at 6 months post procedure | 6 months post procedure
  Proportion of subjects with complete occlusion of the target aneurysm, ≤50% stenosis of the parent artery at the target intracranial aneurysms (IA) at 6 months as assessed by angiography, and in whom an unplanned alternative treatment of the target IA had not been performed within 6 months.
Complete aneurysm occlusion at 6 months post procedure | 6 months post procedure
  Complete occlusion defined as complete obliteration of the aneurysm sac, including the neck (Raymond I).
Retreatment Rate at 6 months and 1 year post procedure | 6 months, 1 year post procedure
  The percentage of target aneurysms that are retreated at any time up to and including the 6 months and 1 year follow-up visit will be evaluated. Retreatment will be defined as any additional treatment of the target aneurysm after the index procedure (retreatment includes staged procedures), and (regardless of whether retreatment is by surgery or endovascular treatment) due to recanalization, rupture or bleeding.
In-Stent Stenosis at 6 months post procedure | 6 months post procedure
  In-stent stenosis defined as greater than 50% narrowing of the vessel within the stent or within 5mm of either end of the stent.
Modified Rankin Scale (mRS) at 30 days, 6 months and 1 year post procedure | 30 days, 6 months, 1 year post procedure
  Observed scores on the Modified Rankin Scale will be presented at baseline (pre-procedure) and follow-up (30 days, 6 and 12 months post-procedure). The number and percentage of subjects who have an mRS ≤ 2 will be evaluated.
Major ipsilateral stroke at 30 days, 6 months and 1 year post procedure | 30 days, 6 months, 1 year post procedure
  National Institute of Health Stroke Scale (NIHSS) was used to assess patients after stroke in an 11-item scale with potential scores ranging from 0 to 42. Higher values represent a worse outcome. A major stroke is defined as a new neurological event which is ipsilateral and in the vascular distribution territory of the stenting procedure and that results in an increase of ≥ 4 on the NIHSS as compared to baseline.
All-cause mortality at 30 days, 6 months and 1 year post procedure | 30 days, 180 days and 1 year post procedure
  Deaths due to any cause are calculated.
Incidence of adverse events/serious adverse events during 30 days, 6 months and 1 year post procedure | 30 days, 6 months and 1 year post procedure
  Percentage (%) of participants who experienced adverse events/serious adverse events.
In-stent thrombosis at 6 months post procedure | 6 months post procedure
  Stent thrombosis defined as a thrombotic occlusion of a stent.
Rate of Device defect | within 1 year of whole trial
  Device defects refer to the unreasonable risks that may endanger human health and life safety during the normal use of medical devices in the course of clinical trials, such as label errors, quality problems, failures, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxin Yang, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China